CLINICAL TRIAL: NCT03959150
Title: A Multi-center, II Phase，Randomized Controlled Clinical Study of Capecitabine Metronomic Chemotherapy After Gemcitabine Plus Capecitabine Standard Adjuvant Therapy for Stage II/III Pancreatic Cancer
Brief Title: Metronomic Chemotherapy With Capecitabine for Pancreatic Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jun Zhang, Chair of Department of Oncology, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Metro-PC
Record Dates: First submitted 2019-05-18; First posted 2019-05-22 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Capecitabine metronomic chemotherapy (Experimental): Capecitabine 500mg/m2 po qd
  Interventions: Drug: Capecitabine
- Observation (No Intervention): Observation

INTERVENTIONS:
Drug: Capecitabine — Oral fluorouracil
  Other Names: Xeloda
  Arms: Capecitabine metronomic chemotherapy

SUMMARY:
The latest guidelines recommend Gemcitabine plus Capecitabine as the first choice of adjuvant chemotherapy for pancreatic cancer patients in good physical condition. In order to prolong the survival of patients and improve the cure rate, metronomic chemotherapy with capecitabine is a safe, effective and economical treatment mode after adjuvant chemotherapy. This study is trying to determine that compared with observation group, if capecitabine metronomic medication is a better choice after adjuvant chemotherapy.

DETAILED DESCRIPTION:
Capecitabine (Xeloda ®) is currently the most biologically active oral fluoropyrimidine drug, and is widely used in adjuvant therapy for pancreatic cancer. It is usually taken twice a day (in the morning and in the evening) for 2 weeks, followed by a 1 week break before repeating the next dosage cycle. In this study, capecitabine will be prescribed as dosage of 500mg/m2, and maintain for a whole year after the standard treatment in stage II/III pancreatic cancer patients. 1 year disease-free survival is set as the primary outcome, OS, RFS, AEs and exploratory biomarkers including effects of metronome chemotherapy on immune cells, such as NK cells, T cells, TAMs, B cells, etc are also observed as the secondary outcomes. Statistical analysis are made to see compared with observation group, whether this metronomic therapy of capecitabine ( 500mg/m2) will bring benefit to pancreatic cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed pancreatic invasive ductal adenocarcinoma.
2. The patient underwent surgery for pancreatic tumor resection, and no gross residual lesions were found postoperatively (R2).
3. Stage II/III pancreatic cancer was determined according to AJCC/UICC TNM stage eighth.
4. At least 6 cycles of gemcitabine plus capecitabine chemotherapy have been completed.
5. Age 18-70 years old, gender not limited.
6. ECOG performance score is 0 or 1.
7. Without dysphagia, able to tolerate oral administration.
8. No relevant clinical or imaging evidence of recurrence or metastasis showing within the 28 days before random.
9. Chemotherapy with capecitabine combined with gemcitabine regimen was given within 12 weeks after surgery, and last chemotherapy to random time ≤ 6 weeks.
10. Adequate bone marrow, liver, and kidney function in measurements taken within 7 days before registration ：
11. Hemoglobin ≥ 90 g/L, Platelet count ≥ 100×109/L, Absolute granulocyte count ≥ 1.5×109/L.

    i. Note: patients should not receive blood transfusion or growth factor support within 14 days before collection of blood samples.
12. Serum creatinine≤ 1.5 ULN, and calculated creatinine clearance of ≥ 60 mL/min/1.73m2.
13. AST and ALT ≤ 2.5 X ULN, serum total bilirubin ≤ 1.5 X ULN (Patients with Gilbert syndrome with total bilirubin≤ 3 X ULN can be enrolled).
14. INR or PT ≤ 1.5×ULN，unless the patient is receiving anticoagulant therapy and the PT value is within the expected therapeutic range of the anticoagulant.
15. Electrocardiogram and cardiac function were not contraindicated in chemotherapy.
16. Women should have a negative pregnancy test, and all the patients have no planning within 3 years and should take contraceptive measures during treatment.
17. Informed consent form signed.

Exclusion Criteria:

1. Other pathological types of pancreatic malignancies (e.g. neuroendocrine carcinoma, large cell carcinoma, signet ring cell carcinoma, etc.).
2. With distant metastasis or malignant pleural effusion.
3. Pregnant and breast-feeding women.
4. Unable to oral medication.
5. Previous or concurrent malignancies, excluding curatively treated in situ carcinoma of the cervix or non-melanoma skin cancer, unless at least 5 years have elapsed since last treatment and the patient is considered cured.
6. A history of transient ischemic attack, cerebrovascular accident, thrombosis, or thromboembolism (pulmonary embolism or deep venous thrombosis) within 180 days before randomization.
7. Any of the following uncontrolled or severe cardiovascular disease history:
8. Myocardial infarction occurred 180 days before randomization.
9. Uncontrolled angina occurred within 180 days before randomization.
10. Heart failure of class III or IV (according to New York Heart Association functional classification).
11. Uncontrolled hypertension after appropriate treatment (e.g. Systolic blood pressure ≥150mmHg or diastolic blood pressure ≥90mmHg for 24h or longer).
12. Arrhythmias that require treatment, including pacemakers.
13. Serious drug allergy.
14. Uncontrolled diabetes or systemic infection.
15. Known dihydro pyrimidine dehydrogenase (DPD) deficiency.
16. Any other reasons the investigator considers the patient should not participate in the study.
17. Without personal freedom and independent civil capacity.
18. Already enrolled into other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Estimated)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
One year disease-free survival | 1 year
  was defined as the rate of disease recurrence, metastasis or death due to disease progression within 1 year after the surgery

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 year
  was defined as the time from the date of surgery until the date of any death occurred
Recurrence-free Survival (RFS) | 1 year
  was defined as the time from the date of surgery until the date of local recurrence of the tumor
AEs | 5 year
  Hand and foot syndrome and other treatment related AE
Exploratory biomarkers | 1 yaer
  including effects of metronome chemotherapy on immune cells, such as NK cells, T cells, TAMs, B cells, etc

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD & Ph. D, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siravegna G, Bardelli A. Blood circulating tumor DNA for non-invasive genotyping of colon cancer patients. Mol Oncol. 2016 Mar;10(3):475-80. doi: 10.1016/j.molonc.2015.12.005. Epub 2015 Dec 17. PMID 26774880
- [Background] Witkowski ER, Smith JK, Tseng JF. Outcomes following resection of pancreatic cancer. J Surg Oncol. 2013 Jan;107(1):97-103. doi: 10.1002/jso.23267. Epub 2012 Sep 18. PMID 22991309
- [Background] Ansari D, Gustafsson A, Andersson R. Update on the management of pancreatic cancer: surgery is not enough. World J Gastroenterol. 2015 Mar 21;21(11):3157-65. doi: 10.3748/wjg.v21.i11.3157. PMID 25805920
- [Background] Liao WC, Chien KL, Lin YL, Wu MS, Lin JT, Wang HP, Tu YK. Adjuvant treatments for resected pancreatic adenocarcinoma: a systematic review and network meta-analysis. Lancet Oncol. 2013 Oct;14(11):1095-1103. doi: 10.1016/S1470-2045(13)70388-7. Epub 2013 Sep 12. PMID 24035532
- [Background] Ferrone CR, Pieretti-Vanmarcke R, Bloom JP, Zheng H, Szymonifka J, Wargo JA, Thayer SP, Lauwers GY, Deshpande V, Mino-Kenudson M, Fernandez-del Castillo C, Lillemoe KD, Warshaw AL. Pancreatic ductal adenocarcinoma: long-term survival does not equal cure. Surgery. 2012 Sep;152(3 Suppl 1):S43-9. doi: 10.1016/j.surg.2012.05.020. Epub 2012 Jul 3. PMID 22763261
- [Background] Narang AK, Miller RC, Hsu CC, Bhatia S, Pawlik TM, Laheru D, Hruban RH, Zhou J, Winter JM, Haddock MG, Donohue JH, Schulick RD, Wolfgang CL, Cameron JL, Herman JM. Evaluation of adjuvant chemoradiation therapy for ampullary adenocarcinoma: the Johns Hopkins Hospital-Mayo Clinic collaborative study. Radiat Oncol. 2011 Sep 28;6:126. doi: 10.1186/1748-717X-6-126. PMID 21951377
- [Background] Kalser MH, Ellenberg SS. Pancreatic cancer. Adjuvant combined radiation and chemotherapy following curative resection. Arch Surg. 1985 Aug;120(8):899-903. doi: 10.1001/archsurg.1985.01390320023003. PMID 4015380
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Javle M, Hsueh CT. Updates in Gastrointestinal Oncology - insights from the 2008 44th annual meeting of the American Society of Clinical Oncology. J Hematol Oncol. 2009 Feb 23;2:9. doi: 10.1186/1756-8722-2-9. PMID 19236713
- [Background] Oettle H, Neuhaus P, Hochhaus A, Hartmann JT, Gellert K, Ridwelski K, Niedergethmann M, Zulke C, Fahlke J, Arning MB, Sinn M, Hinke A, Riess H. Adjuvant chemotherapy with gemcitabine and long-term outcomes among patients with resected pancreatic cancer: the CONKO-001 randomized trial. JAMA. 2013 Oct 9;310(14):1473-81. doi: 10.1001/jama.2013.279201. PMID 24104372
- [Background] Uesaka K, Boku N, Fukutomi A, Okamura Y, Konishi M, Matsumoto I, Kaneoka Y, Shimizu Y, Nakamori S, Sakamoto H, Morinaga S, Kainuma O, Imai K, Sata N, Hishinuma S, Ojima H, Yamaguchi R, Hirano S, Sudo T, Ohashi Y; JASPAC 01 Study Group. Adjuvant chemotherapy of S-1 versus gemcitabine for resected pancreatic cancer: a phase 3, open-label, randomised, non-inferiority trial (JASPAC 01). Lancet. 2016 Jul 16;388(10041):248-57. doi: 10.1016/S0140-6736(16)30583-9. Epub 2016 Jun 2. PMID 27265347
- [Background] Neoptolemos JP, Moore MJ, Cox TF, Valle JW, Palmer DH, McDonald AC, Carter R, Tebbutt NC, Dervenis C, Smith D, Glimelius B, Charnley RM, Lacaine F, Scarfe AG, Middleton MR, Anthoney A, Ghaneh P, Halloran CM, Lerch MM, Olah A, Rawcliffe CL, Verbeke CS, Campbell F, Buchler MW; European Study Group for Pancreatic Cancer. Effect of adjuvant chemotherapy with fluorouracil plus folinic acid or gemcitabine vs observation on survival in patients with resected periampullary adenocarcinoma: the ESPAC-3 periampullary cancer randomized trial. JAMA. 2012 Jul 11;308(2):147-56. doi: 10.1001/jama.2012.7352. PMID 22782416
- [Background] Neoptolemos JP, Palmer DH, Ghaneh P, Psarelli EE, Valle JW, Halloran CM, Faluyi O, O'Reilly DA, Cunningham D, Wadsley J, Darby S, Meyer T, Gillmore R, Anthoney A, Lind P, Glimelius B, Falk S, Izbicki JR, Middleton GW, Cummins S, Ross PJ, Wasan H, McDonald A, Crosby T, Ma YT, Patel K, Sherriff D, Soomal R, Borg D, Sothi S, Hammel P, Hackert T, Jackson R, Buchler MW; European Study Group for Pancreatic Cancer. Comparison of adjuvant gemcitabine and capecitabine with gemcitabine monotherapy in patients with resected pancreatic cancer (ESPAC-4): a multicentre, open-label, randomised, phase 3 trial. Lancet. 2017 Mar 11;389(10073):1011-1024. doi: 10.1016/S0140-6736(16)32409-6. Epub 2017 Jan 25. PMID 28129987
- [Background] Khorana AA, Mangu PB, Berlin J, Engebretson A, Hong TS, Maitra A, Mohile SG, Mumber M, Schulick R, Shapiro M, Urba S, Zeh HJ, Katz MHG. Potentially Curable Pancreatic Cancer: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2017 Jul 10;35(20):2324-2328. doi: 10.1200/JCO.2017.72.4948. Epub 2017 Apr 11. PMID 28398845